CLINICAL TRIAL: NCT05598515
Title: Single Arm Prospective Trial of Time-restricted Feeding to Reduce Inflammation in Fanconi Anemia
Brief Title: Time-restricted Feeding to Reduce Inflammation in Fanconi Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-0751
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Fanconi Anemia
MeSH Terms: conditions — Fanconi Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Time-Restricted Feeding (Experimental)
  Interventions: Behavioral: Time-Restricted Feeding

INTERVENTIONS:
Behavioral: Time-Restricted Feeding — Participants will be asked to eat for only 8 hours out of 24 hours in a day.

SUMMARY:
The main reason for this research study is to determine whether time-restricted eating will reduce inflammation in the bodies of persons with Fanconi anemia (FA) and whether time-restricted eating will improve function in people with FA and neurological changes. Participants will be asked to eat for only 8 hours out of 24 hours in a day.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FA with neuroinflammation
* Age ≥ 12 years old

Exclusion Criteria:

* None

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with neuroinflammation | 6 months
  Presence of neuroinflammation will be measured with a clinical head MRI

CONTACTS AND LOCATIONS:
Overall Officials: Stella Davies, MBBS, PhD, MRCP, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States